CLINICAL TRIAL: NCT03683303
Title: The Mobile Applications (APP) for Patient Education Has Promoted the Knowledge, Skills on the Wound Care and Reduced the Anxiety of Wound Care
Brief Title: The Effects of Educational Program Using APP on Pre-Discharge Knowledge, Skills and Anxiety of Wound Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: KMUHIRB-E(II)-20160030
Record Dates: First submitted 2018-09-17; First posted 2018-09-25 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Wound
MeSH Terms: conditions — Wounds and Injuries | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mobile applications (APP) (Experimental): A total of 70 participants were randomized to each group for 35 people, the control group receiving the oral patient education and the experimental group receiving patient education using mobile applications. Both groups collected data using "Wound Care Knowledge Scale," "Wound Care Skills Scale," "State Trait Anxiety Inventory" and "Heart Rate Variability" at three phases, including before the intervention (T1), after 3 times of intervention (T2), and before discharge from hospital (T3).
  Interventions: Behavioral: mobile applications (APP)
- oral education (Active Comparator): A total of 70 participants were randomized to each group for 35 people, the control group receiving the oral patient education and the experimental group receiving patient education using mobile applications. Both groups collected data using "Wound Care Knowledge Scale," "Wound Care Skills Scale," "State Trait Anxiety Inventory" and "Heart Rate Variability" at three phases, including before the intervention (T1), after 3 times of intervention (T2), and before discharge from hospital (T3).
  Interventions: Behavioral: oral education

INTERVENTIONS:
Behavioral: mobile applications (APP) — the experimental group receiving education using Mobile Application (APP), collected data using "Wound Care Knowledge Scale," "Wound Care Skills Scale," "State Trait Anxiety Inventory" and "Heart Rate Variability" at three phases, including before the intervention (T1), after 3 times of intervention (T2), and before discharge from hospital (T3). The SPSS 22.0 for Windows was used for statistics analyses.
  Arms: mobile applications (APP)
Behavioral: oral education — the control group receiving the oral education, collected data using "Wound Care Knowledge Scale," "Wound Care Skills Scale," "State Trait Anxiety Inventory" and "Heart Rate Variability" at three phases, including before the intervention (T1), after 3 times of intervention (T2), and before discharge from hospital (T3).
  Arms: oral education

SUMMARY:
The purposes of this study were to understand the effects of mhealth App on wound care knowledge, wound care skills, and anxiety related to dressing change when compared to traditional health education before patients discharged from hospital.

DETAILED DESCRIPTION:
1. Research design:

   This study employed a single-blind experimental design. Study participants were randomized into the experimental and control groups. Participants in the experimental group used the mHealth App as intervention while those in the control group received normal verbal instructions. The levels of wound care knowledge, skills, and anxiety related to dressing change in the two groups were compared before intervention (T1), after intervention (T2), and before discharge (T3).
2. Study setting & samples:

The recruitment site of this study was conducted in a plastic surgery ward at a 1500-bed university hospital located in Southern of Taiwan. Samples were recruited either hospitalized patients or their primary caregivers from March to December 2016. Inclusion criteria were of Taiwanese nationality, were aged 20 years and above, had a wound classification score of 6-10 points according to Strauss (2000), required self-care of wound at home, and had a habit of using smartphones. Exclusion criteria included special care conditions, such as (1) other comorbidities (such as severe infection or severe compression injuries with comorbid open fractures) and (2) being a special patient, such as one with mental illness. Sample estimation based on the F test of MANOVA statistics was carried out using the G Power 3.1 software. Each group had at least 31 samples (effect size = 0.25, ∝ = 0.05, power = 0.85). A total of 76 participants satisfied the inclusion criteria for this study. There were 6 patients who were not willing to participate in this study; therefore, 35 participants were randomized enrolled in each of the experimental and control groups.

ELIGIBILITY:
Inclusion Criteria:

* aged 20 years and above.
* wound classification score of 6-10 points according to Strauss (2000).
* required wound self-care at home or care by their primary caregivers.
* had a habit of using smartphones.

Exclusion Criteria:

* other comorbidities (such as severe infection or severe compression injuries with comorbid open fractures).
* being a special patient, such as one with mental illness.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
wound care knowledge | 20 minutes
  wound care knowledge scale was designed by Li (2008) and was used in the studies of Shao (2013) and Liu (2016). The content validity index (CVI) of this 20-item scale was 1.00 for its feasibility, 0.94 for its definiteness and 0.98 for its Appropriateness. A higher score indicates the higher level of wound care knowledge.

SECONDARY OUTCOMES:
wound care skills | 30 minutes
  wound care skills scale was designed by Chen (2010) with 11 items. The CVI for each item was between 0.8 and 1.0 with good validity. The internal consistency reliability of this scale (Cronbach's α) was 0.87. A higher score indicates the higher level of wound care skills. This scale was assessed by healthcare professionals when patients or their caregivers performed wound dressing change.
wound care anxiety | 20 minutes
  State-Trait Anxiety Inventory (STAI) was designed by Spielberger, Gorsuch, & Lushene (1970) with 20 items for assessing trait anxiety and 20 for state anxiety. The internal consistency reliability for the scale have ranged from .86 to .95 and test-retest reliability have ranged from .65 to .75 over a 2-month interval (Spielberger et al., 1983). The revised Chinese version of the STAI scale was 0.9 for situation-specific anxiety and 0.86 for trait anxiety (Chung & Lung, 1984). A higher score indicates the higher level of wound care anxiety.
Heart rate variability (HRV) | 10 minutes
  Heart rate variability (HRV) was measured by the ANS Watch (Department of Health Medical Device Permit Numbers: 001525) to record the variation in the time interval between heartbeats. It can indicate the levels of anxiety from the inputs of the sympathetic and the parasympathetic nervous system and humoral factors. When the level of anxiety is high, patients' physiological effects decreasing in HRV(Huang, Lin, Huang, &Hung, 2008).
Blood pressure(BP) | 10 minutes
  Both systolic blood pressure (SBP) and diastolic blood pressure (DBP) were measured by the ANS Watch (Department of Health Medical Device Permit Numbers: 001525) to record the variation in the time interval between blood pressure. It can indicate the levels of anxiety from the inputs of the sympathetic and the parasympathetic nervous system and humoral factors. When the level of anxiety is high, patients' physiological effects increase in systolic blood pressure (SBP) and diastolic blood pressure (DBP) (Huang, Lin, Huang, &Hung, 2008).
Heart rate (HR) | 10 minutes
  Heart rate was measured by the ANS Watch (Department of Health Medical Device Permit Numbers: 001525) to record the variation in the time interval between heartbeats. It can indicate the levels of anxiety from the inputs of the sympathetic and the parasympathetic nervous system and humoral factors. When the level of anxiety is high, patients' physiological effects increase in heart rate(Huang, Lin, Huang, &Hung, 2008).
High frequency power (HF) | 10 minutes
  High frequency power (HF) was measured by the ANS Watch (Department of Health Medical Device Permit Numbers: 001525) to record the variation in the time interval between heartbeats. It can indicate the levels of anxiety from the inputs of the sympathetic and the parasympathetic nervous system and humoral factors. When the level of anxiety is high, patients' physiological effects decreasing in HF(Huang, Lin, Huang, &Hung, 2008).
Low frequency power (LF) | 10 minutes
  Low frequency power (LF) was measured by the ANS Watch (Department of Health Medical Device Permit Numbers: 001525) to record the variation in the time interval between heartbeats. It can indicate the levels of anxiety from the inputs of the sympathetic and the parasympathetic nervous system and humoral factors. When the level of anxiety is high, patients' physiological effects increase in LF(Huang, Lin, Huang, &Hung, 2008).
The ratio of LF/HF | 10 minutes
  Heart rate variability was measured by the ANS Watch (Department of Health Medical Device Permit Numbers: 001525) to record the variation in the time interval between heartbeats. It can indicate the levels of anxiety from the inputs of the sympathetic and the parasympathetic nervous system and humoral factors. When the level of anxiety is high, patients' physiological effects increase in ratio of LF/HF(Huang, Lin, Huang, &Hung, 2008).

CONTACTS AND LOCATIONS:
Overall Officials: ya-ping 雅萍 Hou 侯, Principal Investigator — Kaohsiung Medical University Chung-Ho Memorial Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chang HY, Hou YP, Yeh FH, Lee SS. The impact of an mHealth app on knowledge, skills and anxiety about dressing changes: A randomized controlled trial. J Adv Nurs. 2020 Apr;76(4):1046-1056. doi: 10.1111/jan.14287. Epub 2019 Dec 20. PMID 31814140